CLINICAL TRIAL: NCT00688675
Title: GERD Segmentation: Document How Swiss GPs Allocate Their GERD Patients to the Three GERD Patient Segments
Brief Title: Gastroesophageal Reflux Disease (GERD) Segmentation: Document How Swiss General Practitioners (GPs) Allocate Their GERD Patients to the Three GERD Patient Segments
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr med Madeleine Billeter, AstraZeneca AG, Switzerland
Other Study IDs: NIS-GCH-NEX-2007/1
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: GERD
Keywords: GERD; Pharmacoepidemiology
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated GERD pts: Previously diagnosed GERD patients on treatment in Switzerland

SUMMARY:
Document how Swiss GPs allocate their GERD patients to the three GERD patient segments (according to King et al.) and how treated GERD patients are affected by their GERD treatment

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed GERD patients
* on treatment for at least 2 weeks

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously diagnosed GERD patients on treatment for at least 2 weeks; in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 2912 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
% patients per GERD patient segment | single visit

SECONDARY OUTCOMES:
Symptom load | single visit
Quality of life | single visit

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Aarau, Switzerland